CLINICAL TRIAL: NCT05673421
Title: Comparison of Exergaming Training With Visual Feedback Training on Upper Limb Functions in Post Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Hafsa Rashid
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Stroke
Keywords: upper limb functions
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Exergaming training
Who Masked: Participant
Masking Description: Visual Feedback Training Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergaming Training Group (Experimental): VR game-assisted intervention will perform for 30-45 min, 5 sessions per week for a duration of 8 weeks.
  Interventions: Other: Exergaming Training
- Visual Feedback Training (Active Comparator): During the visual feedback practices, patients will be seated or in a standing phase close to a table on which a mirror would be placed vertically. The practice would be consisted of nonparetic-side shoulder, elbow, wrist and finger flexion, extension, abduction, adduction movements, task oriented activities like, unscrewing lid of jar ,card stacking, moving coins or marbles from one box to another, Folding towels and stacking them, picking glass, while patient will look into the mirror, -watching the image of their noninvolved hand, thus seeing the reflection of the hand movement projected over the involved hand. After watching the practices on the uninvolved side, patient will be asked to try to do the same movements with the paretic limb while they will be moving the nonparetic limb. Each activity will be performed for 4 min, with a 1 min preparation time between tasks.
  Interventions: Other: Visual Feedback Training

INTERVENTIONS:
Other: Exergaming Training — VR game-assisted intervention will perform for 30-45 min, 5 sessions per week for a duration of 8 weeks
  Arms: Exergaming Training Group
Other: Visual Feedback Training — During the visual feedback practices, patients will be seated or in a standing phase close to a table on which a mirror would be placed vertically. The practice would be consisted of nonparetic-side shoulder, elbow, wrist and finger flexion, extension, abduction, adduction movements, task oriented activities like, unscrewing lid of jar ,card stacking, moving coins or marbles from one box to another, Folding towels and stacking them, picking glass, while patient will look into the mirror, -watching the image of their noninvolved hand, thus seeing the reflection of the hand movement projected over the involved hand. After watching the practices on the uninvolved side, patient will be asked to try to do the same movements with the paretic limb while they will be moving the nonparetic limb.Each activity will be performed for 4 min, with a 1 min preparation time between tasks.
  Arms: Visual Feedback Training

SUMMARY:
Stroke is classically characterized as a neurological deficit attributed to an acute focal injury of the central nervous system (CNS) by a vascular cause, including transient ischemic attack, cerebral infarction, intracerebral hemorrhage, and subarachnoid hemorrhage. It is a major cause of disability and death worldwide. The main purpose of this study to determine the effect of exergaming training compared to visual feedback training on improvement in upper limb function.

DETAILED DESCRIPTION:
Stroke patients have various problems such weight. The loss of motion element involved on ﬁne functions, and the above-mentioned problems can lead to decreased muscle cooperativity of the lower limbs while walking and may also result in an asymmetric gait due to imbalance in the ability to perform exercises. Recent studies on the treatment of stroke patients reported that approaches such as more intensive and repetitive training as compared to conventional general and passive intervention, training related to reality, intervention involving motivation and active participation and forced induction exercise, visual exercise feedback, purpose-oriented training, and task-oriented training are more effective in promoting function after stroke onset. Virtual reality (VR) is frequently used in different disease groups at the clinic for rehabilitation purposes. Xbox Kinect, Nintendo Wii, Sony PlayStation, and Cyber Glove are among the most commonly used VR applications in rehabilitation. Several studies reported that VR applications improved both upper and lower extremity functions and promoted independence in performing activities of daily living.

Games based on virtual reality for stroke rehabilitation are mainly focused on motor rehabilitation. Nevertheless, interest in the integration of cognitive and motor rehabilitation has grown. Research shows that the use of virtual reality-based games improves the range of motion as well as the memory and attention of stroke patients. Benefits of virtual reality games include diverse and intensive exercises, designing exercises tailored to patients' abilities, monitoring patients' progress, and boosting patients' motivation. Game-based virtual reality is an emerging technology in healthcare allowing users to interact with a dynamic 3D environment. Studies show that this technology is an effective, feasible and safe solution which makes rehabilitation more convenient. In addition, computer games increase motivation, satisfaction and involvement of patients.

ELIGIBILITY:
Inclusion Criteria:

* Both genders

  * Subacute and chronic patients of stroke (> 4 weeks).
  * Age: 40-70 years
  * Able to follow verbal instructions related to the visual feedback training.
  * MMSE score >21
  * Modified Ashworth scale (MAS) level 1-3
  * Brunnstrom stages 1-4
  * Fugyl Meyer score limit for upper limb

Exclusion Criteria:

Patients with

* Cognitive and Visual impairments
* Psychological disorder
* History of other neurological disorders
* Pusher's syndrome
* Hemineglect
* Abnormal synergic pattern
* Rheumatoid arthritis or other hand impairments

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Fugyl Meyer Assessment scale | 2 months
  It is now widely used for clinical assessment of motor function. This is an impairment-based test with items organized by sequential recovery stages.
  Change from baseline and 2 months
Box and block test | 2 months
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations, including clients with stroke.
  Change from baseline and 2 months
wolf motor function test | 2 months
  The Wolf Motor Function Test (WMFT) quantifies upper extremity movement ability through timed single- or multiple-joint motions and functional tasks.
  Change from baseline and 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, MSNMPT, Principal Investigator — Riphah International University islamabad
Locations (1):
- Hafsa, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No